CLINICAL TRIAL: NCT05317702
Title: The Duration of Effects of Massage in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Healthy; Pressure Pain Threshold; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderately Painful Massage (Experimental): Participants will be seated in a chair with his or her shirt on. Participants will receive 60 seconds of manual pressure applied to the myofascial trigger point identified in the participant's upper back. The researcher's thumb or index finger will apply a deep manual pressure such that the participant rates the pain = 50/100 on a 101-point numeric pain rating scale with 0 indicating no pain and 100 indicating the most severe pain imaginable. The participant will be asked to rate his or her pain during the massage so the pressure may be adjusted to maintain the 50/100 related pain. Massage will be applied for 60 seconds, 4 times for a total contact time of 240 seconds. During each 30 second break in which manual pressure is released, Pressure Pain Threshold (PPT) to the foot will be examined. PPT will be assessed 2 times immediately after each of the 4 massage applications.
  Interventions: Other: Moderately Painful Massage

INTERVENTIONS:
Other: Moderately Painful Massage — Participants will be seated in a chair with his or her shirt on. Participants will receive 60 seconds of manual pressure applied to the myofascial trigger point identified in the participant's upper back. The researcher's thumb or index finger will apply a deep manual pressure such that the participant rates the pain = 50/100 on a 101-point numeric pain rating scale with 0 indicating no pain and 100 indicating the most severe pain imaginable. The participant will be asked to rate his or her pain during the massage so the pressure may be adjusted to maintain the 50/100 related pain. Massage will be applied for 60 seconds, 4 times for a total contact time of 240 seconds. During each 30 second break in which manual pressure is released, Pressure Pain Threshold (PPT) to the foot will be examined. PPT will be assessed 2 times immediately after each of the 4 massage applications.

SUMMARY:
Massage is a common rehabilitation treatment for musculoskeletal pain. Prior studies indicate massage applied with a deep pressure that induces a moderate amount of pain produces a lessening of pain sensitivity compared to light touch, pain free massage. The investigators now aim to investigate how long pain sensitivity changes last after 4 minutes of moderately painful massage and determine factors that help predict who displays a lessening of pain sensitivity.

ELIGIBILITY:
Inclusion Criteria:

• pain-free

Exclusion Criteria:

* Non-English speaking
* Systemic medical condition known to affect sensation (i.e. uncontrolled diabetes)
* Regular use of prescription pain medication
* Current or history of chronic pain condition
* Currently taking a blood-thinning medication
* Any blood clotting disorder, such as hemophilia
* Contraindications to the application of a blood pressure cuff to the arm, such as: lymphedema or arterial/venous lines
* Contraindications to elevating the arm above the head or exercising the arm with a light weight, such as a recent surgery or fracture
* Investigator is unable to locate myofascial trigger point in the upper trapezius during testing session

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Change in Pressure Pain Threshold | PPT is applied between minutes 1, 2, 3, and 4 of massage. PPT is also applied at minutes 1,3,5,10,15 after massage. A higher PPT indicates a lessening of pain sensitivity.
  A digital pressure algometer will be applied to the web space of the foot opposite the trigger point. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold). Participants will rate the pain experienced during the threshold testing using a 101-point numeric pain rate scale (NPRS) anchored with 0= no pain to 100= the most intense pain sensation imaginable immediately following each testing time.

SECONDARY OUTCOMES:
Temporal Summation | Applied before massage
  Mechanical temporal summation will be examined using a neuropen with neurotip. The neuropen with a neurotip has a semi-sharp point that exerts 40g of pressure. A series of ten pinpricks applied to the palmar surface of the hand opposite the trigger point identified at the beginning of the study visit (if the trigger point is on the left shoulder, the right palm will be used for this test.). Participants will rate the pain intensity of each pinprick using a numerical pain rating scale from 0-100 where 0=no pain and 100=worst pain imaginable. A higher pain rating indicates more pain.
Conditioned Pain Modulation | Applied before massage
  First, PPT will be measured on the foot opposite the trigger point. Second, the arm on the same of the participant's trigger point will be elevated for one minute. A blood pressure cuff will be inflated to 270 mmHg and the participant will return his or her arm to the horizontal position. The participant will repeatedly extend the wrist 20 times with a light weight. Third, PPT will be repeated on the top of the foot.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Wilson, Principal Investigator — UCF
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No